CLINICAL TRIAL: NCT04136756
Title: A Phase 1, Open-label, Multi-center, Dose Escalation and Dose Expansion Study of NKTR-255 in Relapsed or Refractory Hematological Malignancies
Brief Title: NKTR-255 in Relapsed/Refractory Multiple Myeloma & Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-255-02
Record Dates: First submitted 2019-10-09; First posted 2019-10-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Indolent Non-Hodgkin Lymphoma
Keywords: relapsed; refractory; NKTR-255; CAR-T; daratumumab subcutaneous (sc); interleukin-15 (IL-15); MM; NHL; indolent; rituximab; Truxima®
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Recurrence | interventions — NKTR-255; Rituximab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): Evaluation of NKTR-255 as:
  * Monotherapy
  * In combination with daratumumab
  * In combination with rituximab
  This phase will help to determine the RP2D of NKTR-255
  Interventions: Drug: NKTR-255; Drug: Rituximab; Drug: Daratumumab
- Dose Expansion Cohort A (Experimental): Evaluation of RP2D of NKTR-255 as monotherapy in patients with NHL relapsed after CAR-T
  Interventions: Drug: NKTR-255
- Dose Expansion Cohort B (Experimental): Evaluation of RP2D of NKTR-255 as monotherapy and in combination with SC daratumumab in patients with R/R MM
  Interventions: Drug: NKTR-255; Drug: Daratumumab
- Dose Expansion Cohort C (Experimental): Evaluation of RP2D of NKTR-255 as monotherapy and in combination with rituximab in patients with R/R iNHL
  Interventions: Drug: NKTR-255 Q21; Drug: Rituximab

INTERVENTIONS:
Drug: NKTR-255 — NKTR-255 administered by IV infusion every 21 or 28 days to establish safety and tolerability
  Arms: Dose Escalation; Dose Expansion Cohort A; Dose Expansion Cohort B
Drug: NKTR-255 Q21 — NKTR-255 administered by IV infusion every 21 days to establish safety and tolerability
  Arms: Dose Expansion Cohort C
Drug: Rituximab — Rituximab administered intravenously at specified dose on specified days
  Other Names: RITUXAN(R)
  Arms: Dose Escalation; Dose Expansion Cohort C
Drug: Daratumumab — Daratumumab administered subcutaneously at specified dose on specified days
  Other Names: DARZALEX FASPRO(TM)
  Arms: Dose Escalation; Dose Expansion Cohort B

SUMMARY:
Patients will receive intravenous (IV) NKTR-255 in 21 or 28 day treatment cycles. During the Part 1 dose escalation portion of the trial, patients will either receive NKTR-255 as monotherapy, NKTR-255 administered as a doublet with daratumumab subcutaneous (DARZALEX FASPRO TM), or NKTR-255 administered as a doublet with rituximab. After determination of the recommended Phase 2 dose (RP2D) of NKTR-255, NKTR-255 will be evaluated in Part 2. During the Part 2 dose expansion portion of the trial, patients will either receive NKTR-255 as monotherapy, NKTR-255 administered as a doublet with daratumumab subcutaneous (DARZALEX FASPRO TM), or NKTR-255 administered as a doublet with rituximab.

This is a Phase 1 study to evaluate safety and tolerability of NKTR-255 alone and in combination with daratumumab or rituximab.

DETAILED DESCRIPTION:
NKTR-255 is a cytokine that is designed to regulate T and natural killer cell activation, proliferation and promote their anti-tumor effects.

This is a Phase 1, open-label, multi-center, dose escalation, dose expansion, safety follow-up, and survival follow-up of NKTR-255 as a single agent and NKTR-255 in combination with DARZALEX FASPRO TM or rituximab. Study treatment is defined as any investigational treatment(s) or marketed product(s), intended to be administered to a study patient according to the study enrollment.

Part 1 will enroll relapsed/refractory multiple myeloma (MM) and Non-Hodgkin's Lymphoma (NHL) patients. In Part 2, Cohort A will enroll NHL patients who have progressed on a chimeric antigen receptor T-cell (CAR-T) product, Cohort B will enroll MM patients who previously received daratumumab and other anti-CD38 therapies to receive NKTR-255 alone and/or in combination with daratumumab, and Cohort C will enroll indolent Non-Hodgkin's Lymphoma (iNHL) patients who previously received rituximab and other therapies to receive NKTR-255 alone and/or in combination with rituximab.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have relapsed or refractory MM or NHL with no available therapies that would confer clinical benefit for their primary disease.
* For MM patients, measurable relapsed or refractory MM as defined by the IMWG Criteria (Kumar, 2016) following treatment with at least 3 lines of therapy with no other available treatment that would confer benefit.
* For NHL patients, measurable or detectable disease according to International Myeloma Working Group (IMWG) and the Lugano Classification. Extranodal NHL disease that is measurable by fluorodeoxyglucose-positron emission tomography (FDG-PET) imaging only is allowed.
* Estimated glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73 m2.
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2

Patient has the following laboratory test results during Screening:

1. Absolute neutrophil count (ANC) or absolute granulocyte count (AGC) ≥ 1000/µL
2. Platelets ≥ 30,000/µL
3. Hemoglobin ≥ 8g/dL
4. Absolute lymphocytes ≥ 500/µL
5. Leukocytes ≥ 3000/µL

Patients are eligible who also meet all the following criteria in these cohorts of Part 2:

NKTR-255 Monotherapy NHL Group Only:

* Patients with NHL who received a commercially approved CD19 CAR-T product and had PD. The first dose of NKTR-255 will be administered within 30 days of the PD.

NKTR-255 with Daratumumab MM Group Only :

* Patients with MM must have had previous exposure to proteasome inhibitor, immunomodulatory agent (IMiD), and anti-CD38 therapy.
* Patients who previously received daratumumab or other anti-CD38 therapies must have at least 3 months washout.

NKTR-255 with Rituximab Group iNHL Group Only:

* Patients with relapsed or refractory iNHL who previously progressed during or following 1 or more prior systemic rituximab-containing (or another treatment with an anti-CD20 antibody-containing) regimens for lymphoma.

Key Exclusion Criteria:

* Patients who have an active, known, or suspected autoimmune disease.
* Any treatment-related neurotoxicity or cytokine release syndrome (CRS) prior to enrollment into the study should return to baseline before NKTR-255 treatment.
* Active central nervous system (CNS) involvement with NHL.
* Patients who have been previously treated with prior interleukin-2 or interleukin-15.
* Patients who received daratumumab or other anti-CD38 therapies previously must have 3 months washout.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events of NKTR-255 as a single agent | Through study completion, an expected average of 6 months
  Safety and tolerability of NKTR-255 as evaluated by incidence of Dose Limiting Toxicities (DLTs), drug-related Adverse Events (AEs), Serious Adverse Events (SAEs), AEs leading to discontinuation, deaths, clinical laboratory abnormalities per CTCAE v5.
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events of NKTR-255 with daratumumab SC | Through study completion, an expected average of 1 year
  Safety and tolerability of NKTR-255 in combination with daratumumab as evaluated by incidence of drug-related AEs, SAEs, AEs leading to discontinuation, deaths, clinical laboratory abnormalities per CTCAE v5
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events of NKTR-255 with rituximab | Through study completion, an expected average of 1 year
  Safety and tolerability of NKTR-255 in combination with rituximab as evaluated by incidence of drug-related AEs, SAEs, AEs leading to discontinuation, deaths, clinical laboratory abnormalities per CTCAE v5
Evaluate the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of NKTR-255 as a single agent | Through study completion, an expected average of 6 months
Evaluate the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of NKTR-255 in combination with daratumumab SC | Through study completion, an expected average of 1 year
Evaluate the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of NKTR-255 in combination with rituximab | Through study completion, an expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (13):
- United States (13):
  - Western Regional Medical Center - CTCA, Goodyear, Arizona
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Health System, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah N, Perales MA, Turtle CJ, Cairo MS, Cowan AJ, Saeed H, Budde LE, Tan A, Lee Z, Kai K, Marcondes MQ, Zalevsky J, Tagliaferri MA, Patel KK. Phase I study protocol: NKTR-255 as monotherapy or combined with daratumumab or rituximab in hematologic malignancies. Future Oncol. 2021 Sep;17(27):3549-3560. doi: 10.2217/fon-2021-0576. Epub 2021 Jun 22. PMID 34154392
- [Derived] Miyazaki T, Maiti M, Hennessy M, Chang T, Kuo P, Addepalli M, Obalapur P, Sheibani S, Wilczek J, Pena R, Quach P, Cetz J, Moffett A, Tang Y, Kirk P, Huang J, Sheng D, Zhang P, Rubas W, Madakamutil L, Kivimae S, Zalevsky J. NKTR-255, a novel polymer-conjugated rhIL-15 with potent antitumor efficacy. J Immunother Cancer. 2021 May;9(5):e002024. doi: 10.1136/jitc-2020-002024. PMID 34001523